CLINICAL TRIAL: NCT07293754
Title: A Phase 1/2 Trial of RPTR-1-201, a T Cell Receptor Bispecific Therapy, in Advanced Solid Tumors
Brief Title: An Early Phase Trial of RPTR-1-201 in Advanced Solid Tumors
Acronym: RaPTR-101
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Repertoire Immune Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RPTR-1-201-101; 2025-524010-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-03; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Tumor
Keywords: advanced cancer; solid tumors; immunotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): Participants receive RPTR-1-201 at doses and schedules defined by the trial protocol.
  Interventions: Drug: RPTR-1-201
- Combination (Experimental): Participants receive RPTR-1-201 in combination with an approved or investigational PD-1 monoclonal antibody at doses and schedules defined by the trial protocol.
  Interventions: Drug: RPTR-1-201; Drug: PD-1 / PD-L1 monoclonal antibody

INTERVENTIONS:
Drug: RPTR-1-201 — RPTR-1-201
Drug: PD-1 / PD-L1 monoclonal antibody — PD-1/PD-L1 monoclonal antibody
  Arms: Combination

SUMMARY:
This is an early phase trial designed to evaluate the safety, tolerability, and preliminary antitumor activity of RPTR-1-201 in adults with advanced solid tumors. The trial includes dose escalation and dose expansion parts and will evaluate RPTR-1-201 as monotherapy and in combination with an anti-PD-1 monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed locally advanced or metastatic solid tumors that is not amenable to curative treatment.
* At least one measurable lesion per RECIST v1.1 as assessed by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function as defined in the trial protocol.
* Ability to provide written informed consent and comply with trial procedures.

Exclusion Criteria:

* History of another malignancy within 3 years before the first dose of trial intervention, with the exception of malignancies considered cured and not expected to require active therapy (for example, certain skin cancers or in situ malignancies) per protocol.
* Known active leptomeningeal disease or uncontrolled central nervous system metastases.
* Active, clinically significant, autoimmune diseases requiring systemic immunosuppressive therapy.
* Prior allogenic organ transplantation
* Clinically significant uncontrolled medical or psychiatric condition, that in the opinion of the investigator, would increase risk or interfere with trial participation.
* Other protocol-defined inclusion and exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities and treatment-emergent adverse events. | From first dose through 30 days after last dose of trial treatment.
  Number of participants experiencing dose-limiting toxicities and treatment-emergent adverse events, including events considered related to RPTR-1-201, graded according to CTCAE v5.0.
Objective Response Rate (ORR) per RECIST v1.1 | From first dose until end of treatment or documented disease progression, whichever occurs first (assessed up to 24 months).
  Proportion of participants with a best overall response of complete response or partial response per RECIST v1.1, as assessed by the investigator.

SECONDARY OUTCOMES:
Incidence and severity of adverse events and abnormal safety assessments. | From first dose through 30 days after last dose of trial treatment
  Incidence and severity of adverse events, including immune-related adverse events, and abnormal safety assessments (clinical laboratory tests, ECGs, vital signs).
Pharmacokinetics of RPTR-1-201 | First dose until end of treatment (assessed up to 24 months).
  Characterization of the pharmacokinetic maximum observed concentration of RPTR-1-201.
Progression Free Survival (PFS) | From first dose until disease progression, death, or end of trial follow-up, whichever occurs first (assessed up to 24 months).
  Time from first dose of RPTR-1-201 to the earliest date of documented disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Overall survival (OS) | From first dose until death from any cause or end of trial follow-up, whichever occurs first (assessed up to 36 months).
  Time from first dose of RPTR-1-201 to death from any cause.
Time to Response | From first dose until first documented response, disease progression, or end of trial follow-up, whichever occurs first (assessed up to 24 months).
  Time from first dose of RPTR-1-201 to the first documented complete response or partial response per RECIST v1.1.
Pharmacokinetics of RPTR-1-201 (AUC) | First dose until end of treatment (assessed up to 24 months)
  Characterization of the pharmacokinetic area under the curve of RPTR-1-201
Immunogenicity of RPTR-1-201 | First dose until end of treatment (assessed up to 24 months)
  Characterization of the incidence of anti-drug antibodies of RPTR-1-201.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared for this trial.